CLINICAL TRIAL: NCT05047601
Title: A PHASE 2/3, RANDOMIZED, DOUBLE-BLIND, DOUBLE-DUMMY, PLACEBO CONTROLLED STUDY TO EVALUATE THE SAFETY AND EFFICACY OF 2 REGIMENS OF ORALLY ADMINISTERED PF 07321332/RITONAVIR IN PREVENTING SYMPTOMATIC SARS-COV-2 INFECTION IN ADULT HOUSEHOLD CONTACTS OF AN INDIVIDUAL WITH SYMPTOMATIC COVID-19
Brief Title: A Study of a Potential Oral Treatment to Prevent COVID-19 in Adults Who Are Exposed to Household Member(s) With a Confirmed Symptomatic COVID-19 Infection
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C4671006; 2021-002894-24 (EudraCT Number); EPIC-PEP (Other: Alias Study Number)
Record Dates: First submitted 2021-09-01; First posted 2021-09-17 (Actual); Results first posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: COVID-19
Keywords: Severe acute respiratory syndrome coronavirus 2 (SARS-Cov-2)
MeSH Terms: conditions — COVID-19 | interventions — nirmatrelvir; Ritonavir

STUDY DESIGN:
Intervention Model Description: Eligible participants who are asymptomatic household contacts of an individual with symptomatic COVID-19 will be randomized (1:1:1) to receive orally every 12 hours:
  PF-07321332/ritonavir for 5 days followed by placebo for 5 days or PF-07321332/ritonavir for 10 days or Placebo for 10 days
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind Double Dummy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- PF-07321332/ritonavir (5 days) (Experimental): Participants will receive PF-07321332/ritonavir every 12 hours from Day 1 through Day 5 followed by Placebo every 12 hours from Day 6 through Day 10
  Interventions: Drug: PF-07321332; Drug: Placebo for PF-07321332; Drug: Placebo for Ritonavir; Drug: Ritonavir
- PF-07321332/ritonavir (10-Day) (Experimental): Participants will receive PF-07321332/ritonavir every 12 hours from Day 1 through Day 10.
  Interventions: Drug: PF-07321332; Drug: Ritonavir
- Placebo (Placebo Comparator): Participants will receive placebo every 12 hours from Day 1 through Day 10.
  Interventions: Drug: Placebo for PF-07321332; Drug: Placebo for Ritonavir

INTERVENTIONS:
Drug: PF-07321332 — PF-07321332
  Arms: PF-07321332/ritonavir (10-Day); PF-07321332/ritonavir (5 days)
Drug: Placebo for PF-07321332 — Placebo
  Arms: PF-07321332/ritonavir (5 days); Placebo
Drug: Placebo for Ritonavir — Placebo
  Arms: PF-07321332/ritonavir (5 days); Placebo
Drug: Ritonavir — Ritonavir
  Arms: PF-07321332/ritonavir (10-Day); PF-07321332/ritonavir (5 days)

SUMMARY:
The purpose of this clinical trial is to learn whether the study medicine prevent symptoms of COVID-19 in adults who have been exposed to household member(s) with a confirmed symptomatic COVID-19 infection.

All participants in the study will receive treatment for COVID-19 as needed, based on their regular doctor's recommendation. Two-thirds of participants will also receive two study medicines (PF-07321332 and ritonavir) by mouth twice a day for either five or ten days. We will compare the experiences of people receiving the study medicines to those of the people who do not. This will help us determine if the study medicines are safe and effective

ELIGIBILITY:
Inclusion Criteria:

* Participants who have a negative screening SARS-CoV-2 rapid antigen test result and who are asymptomatic household contacts with exposure within 96 hours to an individual who is symptomatic and recently tested positive for SARS CoV-2.
* Fertile participants must agree to use a highly effective method of contraception

Exclusion Criteria:

* History of SARS-CoV-2 infection in the past 6 months
* Experiencing measured fever (documented temperature >38˚C or 100.4˚F) or other signs or symptoms consistent with COVID-19
* Known medical history of active liver disease
* Chronic Kidney Disease or have known moderate to severe renal impairment.
* Known Human Immunodeficiency Virus (HIV) infection with viral load > 400 copies/ml within the last 6 months or taking prohibited medications for HIV treatment
* Suspected or confirmed concurrent active systemic infection
* Active cancer requiring treatment with prohibited medication.
* Current or expected use of any medications or substances that are highly dependent on Cytochrome P450 3A4 (CYP3A4) for clearance or are strong inducers of CYP3A4
* Has received approved, authorized, or investigational anti-SARS-CoV-2 mAb, convalescent plasma, other drugs for treatment of COVID-19, or other anti-SARS-CoV-2 biologic products within 6 months of screening
* Has received any SARS-CoV-2 vaccine within 6 months prior to screening or is expected to receive a SARS-CoV-2 vaccine or other approved, authorized, or investigational postexposure prophylaxis treatments through Day 38.
* Participating in another interventional clinical study with an investigational compound or device, including those for COVID-19
* Known or prior participation in this trial or another trial involving PF-07321332.
* Females who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2954 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2022-04-12 (Actual); Study Completion 2022-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (169):
- United States (64):
  - Cahaba Research Inc, Pelham, Alabama
  - The Institute for Liver Health dba Arizona Clinical Trials, Tucson, Arizona
  - Ascada Health PC, Fullerton, California
  - Optimus Medical Group, San Francisco, California
  - Synergy Healthcare, Bradenton, Florida
  - MOORE Clinical Research, Inc., Brandon, Florida
  - TrueBlue Clinical Research, Brandon, Florida
  - Herco Medical and Research Center Inc, Coral Gables, Florida
  - Advance Clinical Research Group, Cutler Bay, Florida
  - Beautiful Minds Clinical Research Center, Cutler Bay, Florida
  - Qway Research, Hialeah, Florida
  - Eastern Research Inc, Hialeah, Florida
  - Inpatient Research Clinic, Hialeah, Florida
  - Doral Medical Research,LLC, Hialeah, Florida
  - Unlimited Medical Research Group, LLC, Hialeah Gardens, Florida
  - ASCLEPES Research Centers, Lutz, Florida
  - Angels Clinical Research Institute, Miami, Florida
  - LCC Medical Research Institute, LLC, Miami, Florida
  - Premium Medical Research Corp, Miami, Florida
  - Global Health Clinical Trials Corp, Miami, Florida
  - South Florida Research Center, Inc., Miami, Florida
  - University of Miami Health System, Miami, Florida
  - I.V.A.M. Clinical & Investigational Center, LLC, Miami, Florida
  - Medical Research of Westchester Inc, Miami, Florida
  - C'A Research, Miami, Florida
  - ProLive Medical Research, Corp., Miami, Florida
  - Entrust Clinical Research, Miami, Florida
  - Reed Medical Research, Miami, Florida
  - Kendall South Medical Center, Inc., Miami, Florida
  - Clinical Site Partners, Inc dba CSP Miami, Miami, Florida
  - Coral Research Clinic Corp, Miami, Florida
  - Pro-Care Research Center, Corp., Miami Gardens, Florida
  - Savin Medical Group, LLC, Miami Lakes, Florida
  - Omega Research Orlando, Orlando, Florida
  - NAPA Research LLC, Pompano Beach, Florida
  - CDC Research Institute, LLC, Port Saint Lucie, Florida
  - USPA Advance Concept Medical Research Group LLC, South Miami, Florida
  - ASCLEPES Research Centers, Spring Hill, Florida
  - GCP, Global Clinical Professionals, St. Petersburg, Florida
  - Sunrise Research Institute, Sunrise, Florida
  - Santos Research Center, CORP, Tampa, Florida
  - Research by Design, LLC, Chicago, Illinois
  - Accellacare, Ames, Iowa
  - McFarland Clinic, PC, Ames, Iowa
  - Southern Clinical Research Associates. LLC, Metairie, Louisiana
  - Meridian Clinical Research, LLC, Grand Island, Nebraska
  - Quality Clinical Research Inc, Omaha, Nebraska
  - Quality Clinical Research, Omaha, Nebraska
  - Walmart, Las Vegas, Nevada
  - Excel Clinical research, Las Vegas, Nevada
  - Walgreens, Las Vegas, Nevada
  - NYC Health + Hospitals / Harlem, New York, New York
  - Monroe Biomedical Research, Monroe, North Carolina
  - Innovo Research: Wilmington Health, Wilmington, North Carolina
  - PharmaTex Research, LLC, Amarillo, Texas
  - Conroe Willis Medical Research, Conroe, Texas
  - South Texas Clinical Research, Corpus Christi, Texas
  - SingnatureCare Emergency Center, Houston, Texas
  - Trio Clinical Trials, LLC, Houston, Texas
  - C & R Research Services USA, Houston, Texas
  - SMS Clinical Research, LLC, Mesquite, Texas
  - Epic Medical Research, Red Oak, Texas
  - Sun Research Institute, San Antonio, Texas
  - Tranquility Research, Webster, Texas
- Argentina (2):
  - Instituto de Investigaciones Clinicas Zarate, Zárate, Buenos Aires
  - Instituto Médico de la Fundación Estudios Clínicos (Fundación Estudios Clínicos), Rosario, Santa Fe Province
- Brazil (2):
  - Pesquisare Saude S/S Ltda, Santo André, São Paulo
  - Conjunto Hospitalar do Mandaqui, São Paulo
- Bulgaria (17):
  - "Specialized Hospital for Active Treatment of Pneumo-Phthisiatric Diseases-Haskovo" Ltd, Haskovo
  - MHAT "Sv.Ivan. Rilski'' Kozloduy EOOD, Kozloduy
  - Diagnostic-Consultative Center I Lom EOOD, Lom
  - Multiprofile Hospital for Active Treatment- Sveti Nikolay Chudotvoretz EOOD, Lom
  - Medical centre Leo Clinic EOOD, Lovech
  - MHAT Heart and Brain EAD, Pleven
  - DCC Sveti Georgi EOOD, Plovdiv
  - MHAT "St. Panteleimon "- Plovdiv, Plovdiv
  - UMHAT Medica Ruse OOD, Rousse
  - Multiprofile Hospital for Active Treatment - Samokov EOOD, Samokov
  - Multiprofile hospital for active treatment - Sliven to Military Medical Academy, Sliven
  - Diagnostic-Consultative Center XXII- Sofia ЕООD, Sofia
  - UMHATEM N. I. Pirogov EAD, Sofia
  - Specialized hospital for active treatment in pulmonology and phthisiology "Stara Zagora" EOOD, Stara Zagora
  - Medical center Leo Clinic EOOD, Varna
  - MOBAL "D-r Stefan Cherkezov" AD, Veliko Tarnovo
  - Specialized Hospital for Active Treatment of Pneumo-Phthisiatric Diseases Vratsa EOOD, Vratsa
- Colombia (3):
  - Clinica de la Costa LTDA., Barranquilla, Atlántico
  - Caimed S.A.S., Yopal, Casanare Department
  - Cireem Sas, Bogota, Cundinamarca
- Czechia (3):
  - Doktor Brno s.r.o., Brno
  - Zdraví-Fit, s.r.o., Protivín
  - Nemocnice Slany, Slaný
- Medifarma-98 Kft., Nyíregyháza, Hungary
- Japan (5):
  - International University of Health and Welfare Narita Hospital, Narita, Chiba
  - Rakuwakai Otowa Hospital, Kyoto, Kyoto
  - Rinku General Medical Center, Izumisano, Osaka
  - Denenchofu Family Clinic, Ōta-ku, Tokyo
  - Sekino Hospital, Toshimaku, Tokyo
- Hospital Miri, Miri, Sarawak, Malaysia
- Mexico (9):
  - Clinical Research Institute Saltillo S.A. de C.V., Saltillo, Coahuila
  - InfectoLab Consultorios de Especialidad en Infectologia, Tijuana, Estado de Baja California
  - Instituto Jalisciense de Metabolismo, S.C., Guadalajara, Jalisco
  - Christus- Latam Hub Center of Excellence and Innovation Center S.C., Monterrey, Nuevo León
  - Eukarya Pharmasite S.C., Monterrey, Nuevo León
  - EME RED Hospitalaria, Mérida, Yucatán
  - Instituto de Investigaciones Clinicas para la Salud A.C., Durango
  - FAICIC Clinical Research, Veracruz
  - Sociedad de Metabolismo y Corazon S.C., Veracruz
- Centrum Badań Klinicznych Piotr Napora Lekarze Spółka Partnerska, Wroclaw, Poland
- Russia (16):
  - Kirovsk Interdistrict Hospital, Kirovsk, Leningradskaya Oblast'
  - LLC Trekhgorka Medicine, Odintsovo, Moscow Oblast
  - Clinica UZI 4D, Pyatigorsk, Stavropol Kray
  - Barnaul City Hospital Number 5, Barnaul
  - Korolev Medicine, Korolyov
  - KDC "Evromedservis", OJSC, Moscow
  - City Polyclinic #44, Saint Petersburg
  - City Polyclinic No. 109, Saint Petersburg
  - LLC Strategic Medical Systems, Saint Petersburg
  - City Out-patient clinic #112, Saint Petersburg
  - "Research Center Eco-safety" LLC, Saint Petersburg
  - LLC Kurator, Saint Petersburg
  - Saint-Petersburg State Budgetary Healthcare Institution "City Pokrovskaya hospital", Saint Petersburg
  - City Out-patient clinic #4, Saint Petersburg
  - Smolensk State Medical University, Smolensk
  - LLC Family clinic, Yekaterinburg
- South Africa (18):
  - MERC Welkom, Welkom, Free State
  - Worthwhile Clinical Trials, Benoni, Gauteng
  - LCS Clinical Research, Johannesburg, Gauteng
  - Peermed CTC (Pty) Ltd T/A MERC Kempton, Kempton Park, Gauteng
  - Global Clinical Trials, Pretoria, Gauteng
  - Botho Ke Bontle Health Services, Pretoria, Gauteng
  - About Allergy (PTY) Ltd, Pretoria, Gauteng
  - Into Research, Pretoria, Gauteng
  - Clinical Trial Systems (Pty) Ltd, Pretoria, Gauteng
  - Sandton Medical Clinic, Sandton, Gauteng
  - Synapta Clinical Research Center, Durban, KwaZulu-Natal
  - Dr PJ Sebastian Clinical Research Centre, Durban, KwaZulu-Natal
  - Ahmed Al-Kadi Private Hospital, Mayville, Durban, KwaZulu-Natal
  - Limpopo Clinical Research Initiative, Thabazimbi, Limpopo
  - NHC Thohoyandou CRS, Thohoyandou, Limpopo
  - MERC Middelburg, Middelburg, Mpumalanga
  - Madibeng Centre for Research, Brits, North West
  - FCRN Clinical Trial Centre, Vereeniging
- Complexo Hospitalario Universitario da Coruna, A Coruña, Spain
- Thailand (5):
  - The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT),, Pathumwan, Bangkok
  - Faculty of Medicine - Khon Kaen University, Muang, Changwat Khon Kaen
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Faculty of Tropical Medicine, Mahidol University, Bangkok
  - Tropical Medicine Hospital, Bangkok
- Turkey (Türkiye) (7):
  - Ankara University Medical Faculty, Ibni-Sina Hospital, Ankara
  - Istanbul University Istanbul Medical Faculty, Fatih / Istanbul
  - Gaziantep Universitesi Tip Fakultesi Sahinbey Uygulama ve Arastirma Hastanesi, Gaziantep
  - Acibadem University Atakent Hospital, Istanbul
  - Izmir Suat Seren Chest Disease and Surgery Training and Research Hospital, Izmir
  - Mersin University Medical Faculty, Mersin
  - Karadeniz Teknik Universitesi Farabi Hastanesi, Trabzon
- Ukraine (14):
  - Regional Communal Nonprofit Institution "Chernivtsi Regional Clinical Hospital", Chernivtsi
  - Communal non-commercial Enterprise "City Central Clinical Hospital" of Chernivtsi City Council, Chernivtsi
  - Communal non-profit enterprise "City Clinical Hospital #16" of Dnipro City Council, Dnipro
  - Communal nonprofit enterprise "Central City Clinical Hospital of Ivano-Frankivsk City Council", Ivano-Frankivsk
  - Municipal Non-profit Enterprise "Ivano-Frankivsk Regional Phthisiopulmonology Center of, Ivano-Frankivsk
  - Municipal Nonprofit Enterprise "City Student Hospital" of Kharkiv City Council, Kharkiv
  - Municipal Nonprofit Enterprise of Kharkiv Regional Council "Regional Clinical Infectious Diseases, Kharkiv
  - Municipal Nonprofit Enterprise "City Clinic Hospital # 13" of Kharkiv City Council, Kharkiv
  - Polyclinic of Center for Medical Services and Rehabilitation of State Joint-Stock Holding Company, Kyiv
  - Municipal Nonprofit Enterprise "Lviv City Clinic Hospital #4", Lviv
  - Municipal NonProfit Enterprise of the Lviv Regional Council Lviv Regional Information and Analytical, Lviv
  - Municipal Enterprise "Poltava Regional Clinical Infectious Diseases Hospital" of Poltava Regional, Poltava
  - Municipal Enterprise "Volyn Regional Clinical Hospital" of Volyn Regional Council, Tarasove Village
  - Communal Enterprise "Hospital #1" of Zhytomyr City Council, Zhytomyr

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Hammond J, Yunis C, Fountaine RJ, Luscan G, Burr AM, Zhang W, Wisemandle W, Soares H, Baniecki ML, Hendrick VM, Kalfov V, Pypstra R, Rusnak JM. Oral Nirmatrelvir-Ritonavir as Postexposure Prophylaxis for Covid-19. N Engl J Med. 2024 Jul 18;391(3):224-234. doi: 10.1056/NEJMoa2309002. PMID 39018532
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4671006

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who had a negative screening severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) rapid antigen test result and were asymptomatic household contacts of individuals who were symptomatic and recently tested positive for SARS-CoV-2, were included in the study.
Pre-assignment Details: A total of 2880 participants were screened. Out of which, 122 participants were screen failures. 22 participants were not screen failures and were not randomized. 2736 participants were randomized and 2721 participants received study drug.
Groups:
- Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 5 Days: Participants were randomized to receive nirmatrelvir 300 milligrams (mg) and ritonavir 100 mg orally every 12 hours from Day 1 to 5, followed by matching placebo every 12 hours from Day 6 through Day 10.
- Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 10 Days: Participants were randomized to receive nirmatrelvir 300 mg and ritonavir 100 mg orally every 12 hours from Day 1 to 10.
- Placebo: Participants were randomized to receive placebo matched to nirmatrelvir/ritonavir every 12 hours for 10 days from Day 1 through Day 10.
Period: Overall Study
Arm/Group | Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 5 Days | Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 10 Days | Placebo
Started | 921 | 917 | 898
Treated | 913 | 911 | 897
Completed | 877 | 864 | 863
Not Completed | 44 | 53 | 35
Not completed — Lost to Follow-up | 9 | 11 | 7
Not completed — Withdrawal by Subject | 25 | 36 | 23
Not completed — Other | 10 | 6 | 5

BASELINE CHARACTERISTICS:
Population: FAS (Full Analysis Set) included all participants randomly assigned to study intervention regardless of whether or not study intervention was administered.
Groups:
- Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 5 Days: Participants were randomized to receive nirmatrelvir 300 mg and ritonavir 100 mg orally every 12 hours from Day 1 to 5, followed by matching placebo every 12 hours from Day 6 through Day 10.
- Total: Total of all reporting groups
Arm/Group | Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 5 Days | Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 10 Days | Placebo | Total
Number analyzed (Participants) | 921 | 917 | 898 | 2736
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.92 (14.88) | 42.85 (15.02) | 42.39 (14.36) | 43.06 (14.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 502 | 479 | 474 | 1455
  Male | 419 | 438 | 424 | 1281
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 664 | 642 | 643 | 1949
  Not Hispanic or Latino | 257 | 275 | 255 | 787
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 58 | 52 | 49 | 159
  Asian | 8 | 15 | 11 | 34
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 139 | 136 | 132 | 407
  White | 714 | 711 | 704 | 2129
  More than one race | 1 | 1 | 1 | 3
  Unknown or Not Reported | 1 | 2 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Developed Symptomatic RT-PCR or RAT Confirmed SARS-CoV-2 Infection Through Day 14: Among Participants With Negative RT-PCR at Baseline
Description: Percentage of participants who developed symptomatic Reverse Transcriptase Polymerase Chain Reaction (RT-PCR) or Rapid Antigen Test (RAT) confirmed SARS-Cov-2 infection were reported in this outcome measure. Index case was defined as participants with symptomatic COVID-19.
Time Frame: From Day 1 to Day 14
Population: Modified Intent-To-Treat (mITT) population included all participants randomly assigned to study intervention who received at least 1 dose of study intervention and had a negative RT-PCR result at baseline.
Measure: Number; unit: Percentage of participants
Arm/Group | Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 5 Days | Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 10 Days | Placebo
Number analyzed (Participants) | 844 | 830 | 840
Percentage of participants | 2.607 | 2.410 | 3.929
Statistical Analysis 1: Comparison: Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 5 Days vs Placebo; Test type: Superiority; p = 0.1722, Generalized estimating equation (GEE); Model included the fixed effects of treatment, geographic regions and presence of risk factors. Compound symmetry variance-covariance structure; Risk Ratio (RR) = 0.702, 95% CI 2-sided [0.422 to 1.167]
Statistical Analysis 2: Comparison: Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 10 Days vs Placebo; Test type: Superiority; p = 0.1163, GEE; [statistical method as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.645, 95% CI 2-sided [0.373 to 1.115]

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious AEs and AEs Leading to Study and Study Drug Discontinuation
Description: An AE was defined as any untoward medical occurrence in a participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. An SAE was defined as any untoward medical occurrence at any dose that resulted in any of the following outcomes: death; life-threatening ; required inpatient hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity ; congenital anomaly/birth defect; or that was considered as an important medical event. TEAEs were defined as events that started on or after the study medication start date and time. AEs included both serious and all non-serious adverse events. AEs that led to study discontinuation and AEs that led to discontinuation of study intervention and then continued study were also reported in this outcome measure.
Time Frame: From start of study intervention (Day 1) up to end of safety follow-up (Day 38)
Population: Safety analysis set included all participants randomly assigned to study intervention and who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 5 Days | Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 10 Days | Placebo
Number analyzed (Participants) | 912 | 911 | 898
Participants
  TEAEs | 218 | 212 | 195
  SAEs | 3 | 1 | 2
  AEs led to discontinuation of study | 0 | 0 | 0
  AEs led to discontinue study intervention and continued study | 10 | 11 | 14

3. Secondary Outcome: Percentage of Participants Who Developed Symptomatic RT-PCR or RAT Confirmed SARS-CoV-2 Infection Through Day 14: Among Participants With Negative RT-PCR at Baseline With Increased Risk of Severe COVID-19 Illness
Description: Percentage of participants who had a symptomatic RT-PCR or RAT confirmed SARS-Cov-2 infection were reported in this outcome measure. The risk factors associated with severe covid-19 illness included age greater than or equal to 60 years, body mass index greater than 25, social history of smoking and presence of comorbidities. Index case was defined as participants with symptomatic COVID-19.
Time Frame: From Day 1 to Day 14
Population: Modified Intent-To-Treat (mITT2) population included all participants randomly assigned to study intervention who received at least 1 dose of study intervention and had a negative RT-PCR result at baseline and were at increased risk of severe COVID-19 illness.
Measure: Number; unit: Percentage of participants
Arm/Group | Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 5 Days | Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 10 Days | Placebo
Number analyzed (Participants) | 627 | 605 | 606
Percentage of participants | 2.871 | 2.645 | 3.465
Statistical Analysis 1: Comparison: Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 5 Days vs Placebo; Test type: Superiority; p = 0.6766, GEE; Model included the fixed effects of treatment, geographic regions. Compound symmetry variance-covariance structure; Risk Ratio (RR) = 0.880, 95% CI 2-sided [0.484 to 1.602]
Statistical Analysis 2: Comparison: Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 10 Days vs Placebo; Test type: Superiority; p = 0.5070, GEE; Model included the fixed effects of treatment, geographic regions. Compound symmetry variance-covariance structure; Risk Ratio (RR) = 0.809, 95% CI 2-sided [0.433 to 1.512]

4. Secondary Outcome: Percentage of Participants With COVID-19 Related Hospitalization or Death From Any Cause Through Day 28: Among Participants With Negative RT-PCR at Baseline With Increased Risk of Severe COVID-19 Illness
Description: The risk factors associated with severe covid-19 illness included age greater than or equal to 60 years, body mass index greater than 25, social history of smoking and presence of comorbidities.
Time Frame: From Day 1 to Day 28
Population: mITT2 population included all participants randomly assigned to study intervention who received at least 1 dose of study intervention and had a negative RT-PCR result at baseline and were at increased risk of severe COVID-19 illness.
Measure: Number; unit: Percentage of participants
Arm/Group | Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 5 Days | Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 10 Days | Placebo
Number analyzed (Participants) | 627 | 605 | 606
Percentage of participants | 0 | 0 | 0.165

5. Secondary Outcome: Percentage of Participants With Asymptomatic RT-PCR or RAT Confirmed SARS-CoV-2 Infection Through Day 14: Among Participants With Negative RT-PCR at Baseline
Description: Percentage of participants who had asymptomatic RT-PCR or RAT confirmed SARS-CoV-2 infection through day 14 among participants with negative RT-PCR at baseline were reported in this outcome measure. Index case was defined as participants with symptomatic COVID-19.
Time Frame: From Day 1 to Day 14
Population: mITT population included all participants randomly assigned to study intervention who received at least 1 dose of study intervention and had a negative RT-PCR result at baseline.
Measure: Number; unit: Percentage of participants
Arm/Group | Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 5 Days | Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 10 Days | Placebo
Number analyzed (Participants) | 844 | 830 | 840
Percentage of participants | 2.014 | 1.928 | 3.095
Statistical Analysis 1: Comparison: Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 5 Days vs Placebo; Test type: Superiority; p = 0.1869, GEE; [statistical method as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.672, 95% CI 2-sided [0.373 to 1.213]
Statistical Analysis 2: Comparison: Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 10 Days vs Placebo; Test type: Superiority; p = 0.1221, GEE; [statistical method as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.633, 95% CI 2-sided [0.355 to 1.130]

6. Secondary Outcome: Time to RT-PCR or RAT Confirmed SARS-CoV-2 Infection Through Day 14: Among Participants With Negative RT-PCR at Baseline
Description: Number of days between first dose and confirmation of the SARS-CoV-2 infection by RT-PCR or RAT was reported in this outcome measure.
Time Frame: From Day 1 to Day 14
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 5 Days | Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 10 Days | Placebo
Number analyzed (Participants) | 844 | 830 | 840
Days | NA [NA to NA] — Median and the corresponding 95% CI could not be calculated as the proportion of participants who achieved the event were low. | NA [NA to NA] — Median and the corresponding 95% CI could not be calculated as the proportion of participants who achieved the event were low. | NA [NA to NA] — Median and the corresponding 95% CI could not be calculated as the proportion of participants who achieved the event were low.
Statistical Analysis 1: Comparison: Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 5 Days vs Placebo; Test type: Superiority; p = 0.0368, Log Rank
Statistical Analysis 2: Comparison: Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 10 Days vs Placebo; Test type: Superiority; p = 0.0186, Log Rank

7. Secondary Outcome: Percentage of Participants With Symptomatic RT-PCR or RAT Confirmed SARS-CoV-2 Infection Through Day 14: Among Participants With Positive RT-PCR at Baseline
Description: Percentage of participants with a positive RT-PCR result at baseline who had a symptomatic SARS-CoV-2 infection confirmed by RAT or RT-PCR through Day 14 were reported in this outcome measure. Index case was defined as participants with symptomatic COVID-19.
Time Frame: From Day 1 to Day 14
Population: mITT1 population included all participants randomly assigned to study intervention who received at least 1 dose of study intervention and had a positive RT-PCR result at baseline.
Measure: Number; unit: Percentage of participants
Arm/Group | Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 5 Days | Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 10 Days | Placebo
Number analyzed (Participants) | 38 | 48 | 29
Percentage of participants | 28.947 | 45.833 | 37.931
Statistical Analysis 1: Comparison: Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 5 Days vs Placebo; Test type: Superiority; p = 0.4126, GEE; [statistical method as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.750, 95% CI 2-sided [0.378 to 1.491]
Statistical Analysis 2: Comparison: Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 10 Days vs Placebo; Test type: Superiority; p = 0.4273, GEE; [statistical method as in outcome 1, analysis 1]; Risk Ratio (RR) = 1.244, 95% CI 2-sided [0.725 to 2.135]

8. Secondary Outcome: Percentage of Participants With Symptomatic RT-PCR or RAT Confirmed SARS-CoV-2 Infection Through Day 14: Among Participants With Negative, Positive or Missing RT-PCR at Baseline
Description: Percentage of participants with a negative, positive, or missing RT-PCR result at baseline, who had a symptomatic SARS-CoV-2 infection confirmed by RAT or RT-PCR through Day 14 were reported in this outcome measure. Index case was defined as participants with symptomatic COVID-19.
Time Frame: From Day 1 to Day 14
Population: Modified Intent-To-Treat (mITT3) population included all participants randomly assigned to study intervention who received at least 1 dose of study intervention and had a negative, positive or missing RT-PCR result at baseline.
Measure: Number; unit: Percentage of Participants
Arm/Group | Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 5 Days | Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 10 Days | Placebo
Number analyzed (Participants) | 889 | 887 | 873
Percentage of Participants | 3.712 | 4.848 | 5.269
Statistical Analysis 1: Comparison: Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 5 Days vs Placebo; Test type: Superiority; p = 0.1333, GEE; [statistical method as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.726, 95% CI 2-sided [0.478 to 1.103]
Statistical Analysis 2: Comparison: Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 10 Days vs Placebo; Test type: Superiority; p = 0.8088, GEE; [statistical method as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.953, 95% CI 2-sided [0.645 to 1.408]

9. Secondary Outcome: Percentage of Participants With no, Mild, Moderate, or Severe Signs and Symptoms Attributed to COVID-19 Through Day 28: Among Participants With Negative RT-PCR at Baseline
Description: Participants were categorized according to severity of signs and symptoms as no, mild, moderate, severe in this outcome measure. The 12 signs and symptoms included stuffy or runny nose, sore throat, shortness of breath or difficulty breathing, cough, low energy or tiredness, muscle or body aches, headache, chills or shivering, feeling hot or feverish, nausea, vomiting, diarrhea. Participants recorded their daily severity rating of their symptoms over the past 24 hours based on a 4-point scale in which 0 was reported if no symptoms were present; 1 if mild; 2 if moderate; and 3 if severe.
Time Frame: From Day 1 to Day 28
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 5 Days | Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 10 Days | Placebo
Number analyzed (Participants) | 844 | 830 | 840
Percentage of participants
  No | 81.517 | 83.373 | 81.667
  Mild | 7.820 | 8.193 | 7.619
  Moderate | 6.872 | 5.060 | 7.143
  Severe | 2.133 | 2.048 | 2.738
  Missing | 1.659 | 1.325 | 0.833

10. Secondary Outcome: Number of Days of Symptomatic RT-PCR or RAT Confirmed SARS-CoV- 2 Infection Through Day 28: Among Participants With Negative RT-PCR at Baseline
Description: This outcome measure has been reported in terms of number of participants according to days of symptomatic SARS-CoV-2 infection through Day 28.
Time Frame: From Day 1 to Day 28
Population: mITT population included all participants randomly assigned to study intervention who received at least 1 dose of study intervention and had a negative RT-PCR result at baseline. Here, ''Overall Number of Participants Analyzed'' signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 5 Days | Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 10 Days | Placebo
Number analyzed (Participants) | 22 | 20 | 33
Participants
  1 Day of Symptoms | 1 | 7 | 2
  2 Days of Symptoms | 2 | 0 | 1
  3 Days of Symptoms | 0 | 1 | 4
  4 Days of Symptoms | 5 | 0 | 2
  5 Days of Symptoms | 1 | 3 | 3
  6 Days of Symptoms | 0 | 1 | 3
  7 Days of Symptoms | 3 | 4 | 4
  8 Days of Symptoms | 2 | 0 | 5
  9 Days of Symptoms | 0 | 1 | 1
  10 Days of Symptoms | 0 | 0 | 1
  11 Days of Symptoms | 0 | 1 | 1
  12 Days of Symptoms | 2 | 0 | 4
  13 Days of Symptoms | 1 | 1 | 2
  14 Days of Symptoms | 1 | 1 | 0
  18 Days of Symptoms | 2 | 0 | 0
  20 Days of Symptoms | 1 | 0 | 0
  26 Days of Symptoms | 1 | 0 | 0

11. Secondary Outcome: Plasma Concentration Versus Time Summary of Nirmatrelvir (PF-07321332)
Time Frame: Day 1: 1 hour post dose; Day 5: 2 hours pre-dose
Population: Safety analysis set included all participants randomly assigned to study intervention and who received at least 1 dose of study intervention. This outcome measure was not planned to be analyzed for placebo arm. Here, ''Overall Number of Participants Analyzed'' signifies participants evaluable for this outcome measure and ''Number Analyzed'' signifies participants evaluable at specific time points.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 5 Days | Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 10 Days
Number analyzed (Participants) | 476 | 476
Nanograms per milliliter
  Day 1 (1 hour post-dose): number analyzed (Participants) | 159 | 156
  Day 1 (1 hour post-dose) | 1489 (1481.4) | 1472 (1488.2)
  Day 5 (2 hours pre-dose) | 1688 (2093.3) | 1657 (2068.2)

12. Secondary Outcome: Percentage of Participants With Death Event Through Day 38: Among Participants With Negative RT-PCR at Baseline
Description: Percentage of participants with death (all-cause) event were reported in this outcome measure.
Time Frame: From Day 1 to Day 38
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 5 Days | Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 10 Days | Placebo
Number analyzed (Participants) | 844 | 830 | 840
Percentage of participants | 0 | 0 | 0

13. Secondary Outcome: Viral Load in Nasal Samples Over Time: Among Participants With Negative RT-PCR at Baseline
Description: Nasal samples were collected to estimate the viral load in terms of logarithm to base 10 (log10) copies per milliliter in participants with negative RT-PCR at baseline and were reported in this outcome measure.
Time Frame: From Day 1 to Day 14
Population: mITT population included all participants randomly assigned to study intervention who received at least 1 dose of study intervention and had a negative RT-PCR result at baseline. Here 'Number Analyzed' signifies participants evaluable for the specific time points.
Measure: Mean (Standard Deviation); unit: Log 10 copies per milliliter
Arm/Group | Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 5 Days | Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 10 Days | Placebo
Number analyzed (Participants) | 844 | 830 | 840
Log 10 copies per milliliter
  Day 1 | 0.042 (0.265) | 0.035 (0.241) | 0.038 (0.253)
  Day 2: number analyzed (Participants) | 810 | 802 | 809
  Day 2 | 0.078 (0.523) | 0.053 (0.409) | 0.108 (0.611)
  Day 3: number analyzed (Participants) | 823 | 812 | 812
  Day 3 | 0.090 (0.586) | 0.048 (0.374) | 0.147 (0.760)
  Day 4: number analyzed (Participants) | 820 | 808 | 813
  Day 4 | 0.081 (0.537) | 0.057 (0.409) | 0.165 (0.859)
  Day 5: number analyzed (Participants) | 736 | 737 | 742
  Day 5 | 0.079 (0.528) | 0.074 (0.573) | 0.217 (1.063)
  Day 6: number analyzed (Participants) | 817 | 799 | 812
  Day 6 | 0.074 (0.575) | 0.090 (0.670) | 0.189 (0.978)
  Day 7: number analyzed (Participants) | 815 | 798 | 806
  Day 7 | 0.088 (0.586) | 0.053 (0.536) | 0.186 (0.883)
  Day 8: number analyzed (Participants) | 814 | 796 | 805
  Day 8 | 0.096 (0.627) | 0.081 (0.669) | 0.159 (0.860)
  Day 9: number analyzed (Participants) | 810 | 795 | 807
  Day 9 | 0.094 (0.672) | 0.062 (0.596) | 0.135 (0.784)
  Day 10: number analyzed (Participants) | 733 | 715 | 714
  Day 10 | 0.080 (0.616) | 0.064 (0.590) | 0.133 (0.725)
  Day 11: number analyzed (Participants) | 797 | 789 | 793
  Day 11 | 0.103 (0.673) | 0.053 (0.511) | 0.115 (0.707)
  Day 12: number analyzed (Participants) | 803 | 783 | 798
  Day 12 | 0.106 (0.748) | 0.051 (0.447) | 0.103 (0.662)
  Day 13: number analyzed (Participants) | 797 | 791 | 794
  Day 13 | 0.085 (0.642) | 0.052 (0.425) | 0.117 (0.714)
  Day 14: number analyzed (Participants) | 696 | 670 | 686
  Day 14 | 0.108 (0.717) | 0.035 (0.386) | 0.146 (0.798)

14. Secondary Outcome: Viral Load in Nasal Samples Over Time: Among Participants With Positive RT-PCR at Baseline
Description: Nasal samples were collected to estimate the viral load in terms of logarithm to base 10 (log10) copies per milliliter in participants with positive RT-PCR at baseline and were reported in this outcome measure.
Time Frame: From Day 1 to Day 14
Population: mITT1 population included all participants randomly assigned to study intervention who received at least 1 dose of study intervention and had a positive RT-PCR result at baseline. Here 'Number Analyzed' signifies participants evaluable for the specific time points.
Measure: Mean (Standard Deviation); unit: Log 10 copies per milliliter
Arm/Group | Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 5 Days | Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 10 Days | Placebo
Number analyzed (Participants) | 38 | 48 | 29
Log 10 copies per milliliter
  Day 1 | 4.870 (2.041) | 4.470 (1.542) | 4.837 (1.577)
  Day 2: number analyzed (Participants) | 38 | 45 | 28
  Day 2 | 3.286 (2.534) | 2.724 (2.208) | 3.104 (2.909)
  Day 3: number analyzed (Participants) | 38 | 46 | 28
  Day 3 | 2.880 (2.641) | 2.051 (2.212) | 3.255 (2.702)
  Day 4: number analyzed (Participants) | 36 | 47 | 28
  Day 4 | 2.600 (2.427) | 1.514 (2.064) | 2.721 (2.640)
  Day 5: number analyzed (Participants) | 35 | 43 | 27
  Day 5 | 1.470 (2.057) | 1.413 (1.745) | 2.994 (2.677)
  Day 6: number analyzed (Participants) | 38 | 44 | 28
  Day 6 | 1.065 (1.656) | 0.997 (1.696) | 2.466 (2.561)
  Day 7: number analyzed (Participants) | 37 | 45 | 28
  Day 7 | 1.199 (1.747) | 0.913 (1.762) | 1.478 (2.212)
  Day 8: number analyzed (Participants) | 37 | 45 | 28
  Day 8 | 1.212 (1.829) | 0.942 (1.908) | 1.072 (1.663)
  Day 9: number analyzed (Participants) | 38 | 44 | 28
  Day 9 | 1.169 (1.852) | 0.766 (1.858) | 1.103 (1.545)
  Day 10: number analyzed (Participants) | 35 | 45 | 28
  Day 10 | 0.819 (1.656) | 0.541 (1.605) | 0.965 (1.514)
  Day 11: number analyzed (Participants) | 36 | 44 | 28
  Day 11 | 0.623 (1.170) | 0.603 (1.044) | 0.707 (1.116)
  Day 12: number analyzed (Participants) | 37 | 44 | 28
  Day 12 | 0.532 (1.136) | 0.670 (1.204) | 0.436 (0.919)
  Day 13: number analyzed (Participants) | 36 | 45 | 26
  Day 13 | 0.413 (1.098) | 0.313 (1.018) | 0.361 (0.770)
  Day 14: number analyzed (Participants) | 31 | 40 | 25
  Day 14 | 0.284 (1.040) | 0.345 (0.808) | 0.358 (0.735)

15. Secondary Outcome: Number of Days of Hospitalization and Intensive Care Unit (ICU) Stay: Among Participants With Negative RT-PCR at Baseline
Description: This outcome measure has been presented in terms of participants according to number of days of hospitalization and in ICU as 0 days and more than or equal to 1 day.
Time Frame: From Day 1 to Day 28
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 5 Days | Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 10 Days | Placebo
Number analyzed (Participants) | 844 | 830 | 840
Participants
  ICU Visits: 0 Day | 844 | 830 | 840
  ICU Visits: More than or equal to 1 day | 0 | 0 | 0
  Hospitalization Visits: 0 Day | 844 | 830 | 839
  Hospitalization Visits: More than or equal to 1 day | 0 | 0 | 1

16. Secondary Outcome: Number of COVID-19 Related Medical Visits Through Day 28: Among Participants With Negative RT-PCR at Baseline
Description: In this outcome measure number of COVID-19 related medical visits per day were reported. Number of medical visits per day = number of medical visits/number of days follow up through day 28 visit or the last collection date on or before day 28, if day 28 visit was missing.
Time Frame: From Day 1 to Day 28
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Medical visits per day
Arm/Group | Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 5 Days | Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 10 Days | Placebo
Number analyzed (Participants) | 844 | 830 | 840
Medical visits per day | 0.0067 (0.0200) | 0.0057 (0.0201) | 0.0066 (0.0182)
Statistical Analysis 1: Comparison: Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 5 Days vs Placebo; Test type: Superiority; p = 0.7991, Negative binomial regression model; LS Mean Ratio = 0.969, 95% CI 2-sided [0.758 to 1.238]
Statistical Analysis 2: Comparison: Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 10 Days vs Placebo; Test type: Superiority; p = 0.1985, Negative binomial regression model; LS Mean Ratio = 0.847, 95% CI 2-sided [0.657 to 1.091]

ADVERSE EVENTS:
Time Frame: From Day 1 to Day 38
Description: Same event may appear as both SAE and non-SAE but are distinct events. An event may be categorized as serious in 1 participant and non-serious in another, or a participant may have experienced both SAE and non-SAE. Safety population comprised of all participants who received at least 1 dose of study intervention during the study.
Arm/Group | Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 5 Days | Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 10 Days | Placebo
All-Cause Mortality (participants affected / at risk) | 0/912 | 0/911 | 0/898
Serious Adverse Events (participants affected / at risk) | 3/912 | 1/911 | 2/898
Other Adverse Events (participants affected / at risk) | 176/912 | 173/911 | 152/898
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 5 Days (N=912) | Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 10 Days (N=911) | Placebo (N=898)
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 1 | 1 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 5 Days (N=912) | Nirmatrelvir (PF-07321332) 300 mg + Ritonavir 100 mg 10 Days (N=911) | Placebo (N=898)
Diarrhoea (Gastrointestinal disorders) | 23 | 22 | 15
Nausea (Gastrointestinal disorders) | 16 | 12 | 14
Asthenia (General disorders) | 10 | 7 | 17
COVID-19 (Infections and infestations) | 27 | 26 | 36
Nasopharyngitis (Infections and infestations) | 13 | 9 | 6
Upper respiratory tract infection (Infections and infestations) | 20 | 17 | 18
Activated partial thromboplastin time prolonged (Investigations) | 11 | 14 | 22
Alanine aminotransferase increased (Investigations) | 2 | 6 | 11
Blood creatine phosphokinase increased (Investigations) | 12 | 15 | 13
Blood thyroid stimulating hormone increased (Investigations) | 11 | 8 | 10
Fibrin D dimer increased (Investigations) | 18 | 13 | 4
Dysgeusia (Nervous system disorders) | 54 | 62 | 6
Headache (Nervous system disorders) | 15 | 17 | 29
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 2 | 12
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-01-25): https://cdn.clinicaltrials.gov/large-docs/01/NCT05047601/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-15): https://cdn.clinicaltrials.gov/large-docs/01/NCT05047601/SAP_001.pdf